CLINICAL TRIAL: NCT06384417
Title: Adapting an Advance Care Planning Intervention for Use With Patients With Cancer and Their Care Partners: Phase Two
Brief Title: Using an End-of-life Conversation Game to Engage Patients With Cancer in Advance Care Planning: Phase 2
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Lauren Van Scoy, Professor of Medicine, Humanities and Public Health Sciences, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: STUDY00024858
Record Dates: First submitted 2024-04-22; First posted 2024-04-25 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer; Lung Cancer; Genito-Urinary Cancer; Colorectal Cancer; Gastric Cancer; Pancreatic Cancer; Liver Cancer; Head and Neck Cancer; Melanoma
Keywords: Advance Care Planning; Advance Directives; Cancer
MeSH Terms: conditions — Breast Neoplasms; Lung Neoplasms; Urogenital Neoplasms; Colorectal Neoplasms; Stomach Neoplasms; Pancreatic Neoplasms; Liver Neoplasms; Head and Neck Neoplasms; Melanoma; Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hello for Cancer game (Experimental): For this arm, individuals will play the modified Hello game (Hello for Cancer). This game was modified to be better suited for individuals with cancer and their loved ones, and those modifications are now being tested. This game will include questions related to a variety of topics around an individual's cancer experience and medical decision making related to their cancer diagnosis.
  After playing the game, individuals will be asked to reflect on the game questions and provide feedback to inform further modifications.
  Interventions: Behavioral: Hello for Cancer game
- Table Topics game (Placebo Comparator): For this arm, individuals will play commercially available Table Topics game during the research event. This game asks a variety of conversation starting questions, not particularly related to medical decision making.
  Interventions: Other: Table Topics game

INTERVENTIONS:
Behavioral: Hello for Cancer game — To play 'Hello', players are provided 32 open-ended questions in a prearranged order and an equal number of game chips. A player reads aloud the first question. Players then individually write down their answers, and take turns sharing answers with the group (players can opt to pass). Players control how long they share, what they share, and when they are ready to proceed to the next question. During the conversation, players may choose to acknowledge others for a particularly thoughtful, poignant, or even funny comment by giving them a chip. A simple pre-game coin flip determines whether the player with the most chips 'wins' the game ('heads'), or the player with the least amount of chips wins the game ('tails').
  The questions used in Hello for Cancer were modified from the original Hello game based on the results of phase 1 of testing this game in cancer populations. The modifications made to the game will be assessed for acceptability during this study.
  Arms: Hello for Cancer game
Other: Table Topics game — To play Table Topics, players are provided a deck of cards that have a variety of general conversation starter questions. The group takes turns selecting a card and reading it to the group for the group to answer. During the conversation, players may choose to acknowledge others for a particularly thoughtful, poignant, or even funny comment by giving them a chip. A simple pre-game coin flip determines whether the player with the most chips 'wins' the game ('heads'), or the player with the least amount of chips wins the game ('tails').
  Arms: Table Topics game

SUMMARY:
The goal of this clinical trial is to explore feasibility, acceptability, and effectiveness of end-of-life conversation game "Hello" as a tool to help individuals with various solid cancer types (including: breast, gastro-intestinal, lung, melanoma, head and neck, and/or genito-urinary cancers) treated at Penn State Health clinics and their loved ones perform advance care planning (ACP). The main questions it aims to answer are:

What modifications and/or adaptations are necessary to Hello for use in cancer populations?

What impact does participation in Hello event have on health care usage (e.g., number of hospitalizations, ICU admissions, emergency department visits, etc.)? How feasible is it to randomize participants to play either Hello for Cancer or Table Topics?

Participants will:

* Complete pre-game questionnaires
* Play either Hello or Table Topics game
* Complete post-game questionnaires
* Participate in a focus group
* Complete a telephone follow up interview 1-4 months after their event

This study is a continuation of NCT06028152.

DETAILED DESCRIPTION:
Previous studies conducted by the investigators have shown that the Hello game demonstrates successful advance care planning (ACP) engagement in general populations, but has yet to be tailored to meet the unique needs of patients with advanced cancer and their caregivers. Outlining their care preferences by engaging in ACP is an important aspect of care according to patients with advanced cancer. However, only 55% of patients with advanced cancer patients have participated in ACP. These patients have substantial bio-psycho-social stressors that distinguish their ACP needs from others. Tailoring established interventions that foster high quality conversations about medical treatment preferences and end-of-life issues (such as the Hello game) is critically important for this population given its unique needs. As evidenced by qualitative interviews with >200 participants, the Hello game creates a safe environment for sensitive conversations about end-of-life issues and inspired sharing of rich perspectives, with no reported adverse events, excessive burden, or negative emotional effects. That said, the intervention must be adapted for patients with cancer, particularly those with advanced cancer and their caregivers.

Additionally, while several effective ACP interventions exist (including Hello), how best to disseminate these interventions has not been rigorously or systematically studied. In other ongoing and previous studies, the investigators have demonstrated success in both engaging individuals living in underrepresented communities in ACP and successfully enrolling them in interventional research about ACP. The investigators credit these successes to their unique intervention delivery approach called the Community Based Delivery Model (CBDM). The CBDM overcomes key barriers to ACP (such as healthcare distrust, resistance, and hesitancy to discuss end-of-life issues) by leveraging established community connections to recruit participants to participate in ACP interventions as well as research. In the CBDM, trusted community "hosts" (who are leaders from local hospice organizations, senior centers, health agencies) invite participants to attend an ACP event. They introduce the research team to the attendees who may choose to participate in the ACP activity, the research, or both. Hosts are provided with marketing materials and utilize their community network channels to advertise the event. This model allows for research to be conducted more easily within hard to reach and underserved communities such as Black, Hispanic and rural communities- much like the most remote communities across the Penn State Cancer Institute's 28-county catchment area.

Patients with cancer, however, are unique, and may require an alternative approach that involves partnering with their oncology care team to introduce the concept of ACP and encourage participation in ACP and research. Notably, there is evidence that patients are more likely to engage in ACP when recommended by their physician, so how best to approach ACP for cancer patients is unknown. A common approach to ACP intervention research is to use a Healthcare Based Delivery Model (HBDM). In contrast to the CBDM, the HBDM is positioned within the healthcare system (i.e., clinic-based recruitment) as the ACP intervention is recommended by the patient's clinician (rather than through community-based outreach groups). For this intervention delivery approach, research assistants support interactions between clinicians (providers or nurses) to find appropriate patients and garner interest in performing ACP. This model is commonly used to recruit patients for clinical trials, including ACP interventions. For patients with cancer, the HBDM may have some advantages over the CBDM, given the close bonds that form between a patient and clinical care team as they interact frequently during active treatments such as infusions and radiation that often span several hours and weeks. Leveraging these therapeutic relationships may support greater acceptance of opportunities to broach ACP than a community-based model, but this remains unknown.

ELIGIBILITY:
Inclusion Criteria Patient with Cancer:

* Adults (> 18 years old)
* Able to speak and read English and/or Spanish
* Be an individual diagnosed with a solid tumor cancer (e.g., breast, colon, lung, melanoma, head and neck, or genitourinary/prostate cancer) as verified by primary oncologist or is the chosen caregiver for a participant with those cancers
* Receives care at Penn State Health or is the chosen caregiver for a participant treated at Penn State Health

Exclusion Criteria Patient with Cancer:

* Has completed an advance directive since cancer diagnosis as verified by presence in the patient's medical chart
* Has not received treatment for their cancer at a Penn State Health facility in the past year
* Unable to consent to participate in study

Inclusion Criteria Caregiver/Loved one:

* Adults (> 18 years old)
* Able to speak and read English and/or Spanish
* Be the chosen caregiver for a participant with cancer

Exclusion Criteria Caregiver/Loved one:

* Unable to consent to participate in study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-06-27 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Perceptions of modified intervention | immediately post-intervention
  Focus groups will be conducted with individuals randomized to play the Hello for Cancer game. These focus groups will focus on learning about the participants' perception of playing the modified game and identified any questions that need additional modification.
Healthcare Utilization | Baseline to up to two years after participation in research event
  The patient's medical chart will be reviewed to collect data on their medical history as related to their cancer diagnosis. The medical chart will be reviewed for up to two years after participation to capture hospitalizations, intensive care unit admissions, and emergency department visits that occur after the individual's participation in the study.
  Additionally, the patient's chart will be reviewed to identify if since the event any advance directives were uploaded to the medical chart and if there is documentation about conversations regarding medical decision making and ACP with the health care team.

SECONDARY OUTCOMES:
Advance Care Planning Engagement Measure | Baseline
  This 4-item short-version survey measures readiness to perform ACP.
Advance Care Planning Surrogate Decision Maker Engagement Measure | Baseline
  This 17-item survey measures surrogate decision maker readiness to perform ACP.
Satisfaction of Intervention Measure | Immediately post-intervention
  This 8-item survey measures participants' satisfaction with the conversation. Each item is scored on a 1-7 scale with 1 being lowest conversation satisfaction. The items are averaged for the final score ranging 1-7 with 7 indicating the highest conversation satisfaction.
Acceptability of Intervention Measure | Immediately post-intervention
  This 3-item survey measures participants' perceived acceptability of the intervention.
Preliminary efficacy of Hello on ACP behaviors. | Event follow-up interview (one to four months post event)
  During the follow up interview, presence of ACP behaviors since participation in research event will be assessed. Specifically, individuals will be asked if they have completed any advance directives or had conversations with loved ones or family members about advance care planning.

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Van Scoy, MD, Principal Investigator — Penn State College of Medicine
Locations (1):
- Penn State Cancer Institute, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No